CLINICAL TRIAL: NCT03454763
Title: Randomized Phase II Trial in Sstr2 Positive Tumors to Optimize the Interval Between Cycles of PRRT with 177lu-dotatate
Brief Title: Optimizing the Interval Between Cycles of PRRT with 177lu-dotatate in Sstr2 Positive Tumors
Acronym: LUTHREE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Romagnolo per lo Studio dei Tumori Dino Amadori IRST S.r.l. IRCCS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRST100.26
Record Dates: First submitted 2018-02-27; First posted 2018-03-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Neuroendocrine Tumors
Keywords: sst2-positive tumors; Neuroendocrine Tumors; radiolabelled somatostatin analogues (PRRT)
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Intervention Model Description: comparative
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A, Intensive (Experimental): Arm A, Intensive every 5 weeks
  Interventions: Drug: PRRT every 5 weeks
- Arm B, Non Intensive (Experimental): Arm B, Non Intensive every 8-10 weeks
  Interventions: Drug: PRRT every 8-10 weeks

INTERVENTIONS:
Drug: PRRT every 5 weeks — PRRT (radiolabelled somatostatin analogues) every 5 weeks for 5 cycles
  Arms: Arm A, Intensive
Drug: PRRT every 8-10 weeks — PRRT (radiolabelled somatostatin analogues) every 8-10 weeks for 5 cycles
  Arms: Arm B, Non Intensive

SUMMARY:
Randomized Phase II Trial in sstr2 Positive Tumors to Optimize the Interval Between Cycles of PRRT With 177lu-dotatate

DETAILED DESCRIPTION:
The main objective of this randomized phase II comparative study is to evaluate the Progression Free survival (PFS) and the safety as co-primary objective of two different schedule of administrations of 177lu-dotatate: intensive (every 5 weeks) vs no intensive (every 8-10 weeks) The secondary objectives are DCR, the late toxicity, OS and dosimetry. Patients with any tumor histotype documented as sst2-positive in pre-study period will be enrolled in the study.

The study will include a total of 618 planned patients. They will be randomly assigned to receive 5 cycles of PRRT at intervals of 5 or 8-10 weeks between cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Patients must have histologically or cytologically confirmation of neuroendocrine tumors or any other tumor histotype documented as sst2-positive), that may benefit from receptor radionuclide therapy and for which there aren't any other effective treatments. For cerebral sst2-positive tumors, if biopsy is no feasible for technical reason or risk benefit balance, patients may be enrolled if CT or MRI strongly suggest oncological lesion confirming the 68Ga PET-CT dota-peptide SSTr2 positivity..
3. Measurable disease according to RECIST 1.1.criteria also patients without measurable but with evaluable disease disease can be enrolled.
4. Any disease stage is allowed. Patients with documented disease will be admitted to therapeutic phase only if the diagnostic OctreoScan (the tumour uptake will be evaluated with a 3-grade scale, where 1 = liver uptake, 2 > liver uptake and < kidney uptake and 3 > kidney uptake: only tumour uptakes grade 2 and 3 will be considered for therapy) and/or Positron Emission Tomography (PET)/CT 68Ga-peptide images demonstrate a significant uptake in the tumour.
5. Patients with progressive disease in pre-study period (PD within the last 12 months), refractory to conventional standard treatments; clinical progression is allowed
6. Patients with or without concurrent therapy with somatostatin analogs
7. Life expectancy of greater than 6 months.
8. Eastern Cooperative Oncology Group (ECOG) performance status =<2
9. Adequate haematological, liver and renal function: haemoglobin >= 9 g/dL, absolute neutrophil count (ANC) >= 1.5 x 109 /L, platelets >= 100 x 109 /L, bilirubin ≤1.5 X upper normal limit (UNL) , alanine aminotransferase ( ALT) and Aspartate aminotransferase (AST) <2.5 X UNL (< 5 X UNL in presence of liver metastases, creatinine < 2 mg/dL.
10. If female of childbearing potential highly effective birth control methods, according to guideline "Recommendation related to contraception and pregnancy testing in clinical trials", (2014_09_15 section 4.1) are mandatory. Highly effective birth control methods are required beginning at the screening visit and continuing until 6 months following last treatment with study drug. Negative serum pregnancy test for females of childbearing potential within 14 days of starting treatment. Male patient and his female partner who is of childbearing potential must use 2 acceptable methods of birth control (1 of which must include a condom as a barrier method of contraception) starting at screening and continuing throughout the study period and for 6 months after final study drug administration. Two acceptable methods of birth control thus include Condom (barrier method of contraception) and one of the following is required (established use of oral, or injected or implanted hormonal method of contraception by the female partner; placement of an intrauterine device (IUD) or intrauterine system (IUS) by the female partner; additional barrier method like occlusive cap with spermicidal foam/gel/film/cream/suppository in the female partner; tubal ligation in the female partner; vasectomy or other procedure resulting in infertility (eg, bilateral orchiectomy), for more than 6 months.
11. Participant is willing and able to give informed consent for participation in the study.

Exclusion Criteria:

1. Patients treated with chemotherapy and therapeutic radiotherapy within 4 weeks and treated within 2 weeks with palliative radiotherapy, hormonal or biological therapy.
2. Patients treated with previous radiometabolic therapy with an adsorbed dose to the kidney more than 23 Gy and more than 1.8 Gy for the bone marrow or as surrogate of dosimetry (13).
3. Patients which are included in the indication of LUTATHERA®
4. All acute toxic effects of any prior therapy (including surgery radiation therapy, chemotherapy) must have resolved to a grade ≤ 1 according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE)
5. ECOG performance status >2
6. Participation in another clinical trial with any investigational agents within 30 days prior to study screening.
7. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
8. Assessed bone marrow invasion > 50% (with Bone Marrow biopsy or instrumental exams i.e. bone scan or CT or MRI)
9. Pregnant or breastfeeding women are excluded from the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Estimated)
Dates: Start 2016-05-26 (Actual); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
PFS | up to 5 years
  Progression free survival is defined as the time from the randomization date to the date of first observation of documented disease progression or death due to any cause
Incidence of Treatment-Emergent Adverse Events | up to 30 days after last treatment cycle
  The evaluation of Treatment-Emergent Adverse Events, defined as any G3/G4 toxicity from 1st treatment cycle until 30 days after the last treatment cycle will be based on version 4.0 CTC-AE

SECONDARY OUTCOMES:
DCR | up to 5 years
  Disease Control Rate (DCR) is defined as the percentage of patients who have achieved complete response, partial response and stable disease for at least 12 weeks from therapy start. DCR will be evaluated using the new international criteria proposed by the Version 1.1 Response Evaluation Criteria in Solid Tumors (RECIST)
OS | up to 5 years
  Overall Survival (OS) is defined as the time from treatment start to the time of death due to any cause or the date of last contact (censored observation) at the date of data cut-off.

CONTACTS AND LOCATIONS:
Overall Officials: Maddalena Sansovini, MD, Study Chair — IRST IRCCS; Stefano Severi, MD, Principal Investigator — IRST IRCCS
Locations (1):
- Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (IRST), Meldola, FC, Italy

REFERENCES:
- [Derived] Grassi I, Nicolini S, Marini I, Matteucci F, Ranallo N, Di Iorio V, Sarnelli A, Foca F, Monti M, Fabbri L, Fantini L, Rossi A, Paganelli G, Severi S, Sansovini M. Lu-PRRT Used More Intensively on Advanced Gastro-Entero-Pancreatic and Lung Neuroendocrine Neoplasms: Preliminary Results on Toxicity from a Randomized Study. Neuroendocrinology. 2025;115(5):434-445. doi: 10.1159/000542328. Epub 2024 Nov 21. PMID 39571544
- [Derived] Di Franco M, Zanoni L, Fortunati E, Fanti S, Ambrosini V. Radionuclide Theranostics in Neuroendocrine Neoplasms: An Update. Curr Oncol Rep. 2024 May;26(5):538-550. doi: 10.1007/s11912-024-01526-5. Epub 2024 Apr 6. PMID 38581469
- [Derived] Lechner M, Takahashi Y, Turri-Zanoni M, Liu J, Counsell N, Hermsen M, Kaur RP, Zhao T, Ramanathan M Jr, Schartinger VH, Emanuel O, Helman S, Varghese J, Dudas J, Riechelmann H, Sprung S, Haybaeck J, Howard D, Engel NW, Stewart S, Brooks L, Pickles JC, Jacques TS, Fenton TR, Williams L, Vaz FM, O'Flynn P, Stimpson P, Wang S, Hannan SA, Unadkat S, Hughes J, Dwivedi R, Forde CT, Randhawa P, Gane S, Joseph J, Andrews PJ, Royle G, Franchi A, Maragliano R, Battocchio S, Bewicke-Copley H, Pipinikas C, Webster A, Thirlwell C, Ho D, Teschendorff A, Zhu T, Steele CD, Pillay N, Vanhaesebroeck B, Mohyeldin A, Fernandez-Miranda J, Park KW, Le QT, West RB, Saade R, Manes RP, Omay SB, Vining EM, Judson BL, Yarbrough WG, Sansovini M, Silvia N, Grassi I, Bongiovanni A, Capper D, Schuller U, Thavaraj S, Sandison A, Surda P, Hopkins C, Ferrari M, Mattavelli D, Rampinelli V, Facchetti F, Nicolai P, Bossi P, Henriquez OA, Magliocca K, Solares CA, Wise SK, Llorente JL, Patel ZM, Nayak JV, Hwang PH, Lacy PD, Woods R, O'Neill JP, Jay A, Carnell D, Forster MD, Ishii M, London NR Jr, Bell DM, Gallia GL, Castelnuovo P, Severi S, Lund VJ, Hanna EY. Clinical outcomes, Kadish-INSICA staging and therapeutic targeting of somatostatin receptor 2 in olfactory neuroblastoma. Eur J Cancer. 2022 Feb;162:221-236. doi: 10.1016/j.ejca.2021.09.046. Epub 2021 Dec 31. PMID 34980502